CLINICAL TRIAL: NCT03796975
Title: Efficacy of Pioglitazone Hydrochloride and Metformin Hydrochloride Tablets on the Patients With Newly Diagnosed Type 2 Diabetes Mellitus Combined With Non-alcoholic Fatty Liver Disease：an Multicenter，Randomized, Double-blind, Parallel- Controlled Study.
Brief Title: Efficacy of Pioglitazone Hydrochloride and Metformin Hydrochloride Tablets on the Patients With Newly Diagnosed Type 2 Diabetes Mellitus Combined With Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Second Affiliated Hospital of Xi'an Jiaotong University (Other); Shaanxi Aerospace Hospital (Unknown); Genertec Universal Xi'an Aero-Engine hospital (Xi' an) Co., Ltd (Unknown); Xi'an Gaoxin Hospital (Other); Chang'An Hospital (Other); Yan'an people's Hospital (Unknown); Shangluo Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY20172053-1
Record Dates: First submitted 2018-11-11; First posted 2019-01-08 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Type 2 Diabetes Mellitus; Non-alcoholic Fatty Liver Disease; Efficacy
Keywords: Type 2 Diabetes Mellitus; Pioglitazone Hydrochloride and Metformin Hydrochloride Tablets; Randomized Controlled Trial; Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of Pioglitazone and Metformin Tablets (Experimental): dosage form: tablet; dosage:15mg/500mg; frequency: the dose in week 1 is 15mg/500mg, once a day, increased to 15mg/500mg in the second week, twice a day and maintain this dose to 24 weeks duration: 24 weeks; type: oral;
  Interventions: Drug: Combination of Pioglitazone and Metformin Tablets
- Metformin Hydrochloride Tablets (Active Comparator): dosage form: tablet; dosage: 850mg; frequency: the dose in week 1 is 850mg, once a day, increased to 850mg in the second week, twice a day and maintain this dose to 24 weeks duration: 24 weeks; type: oral;
  Interventions: Drug: Metformin Hydrochloride Tablets

INTERVENTIONS:
Drug: Combination of Pioglitazone and Metformin Tablets — 15mg/500mg, oral, 2/day
  Other Names: ka shuang ping
  Arms: Combination of Pioglitazone and Metformin Tablets
Drug: Metformin Hydrochloride Tablets — Oral metformin 850mg, 2/day in the control group
  Other Names: ge hua zhi
  Arms: Metformin Hydrochloride Tablets

SUMMARY:
This is an multicenter, randomized, double-blind, parallel-controlled study to evaluated the efficacy of pioglitazone hydrochloride and metformin hydrochloride tablets on the patients with newly diagnosed type 2 diabetes mellitus combined with non-alcoholic fatty liver disease.

DETAILED DESCRIPTION:
Taking metformin monotherapy as a control, we evaluated the efficacy of pioglitazone hydrochloride and metformin hydrochloride tablets on hepatic fat ultrasound and liver enzyme levels, and observed whether the drug can improve fatty liver in patients with newly diagnosed type 2 diabetes combined with non-alcoholic fatty liver disease. This is an multicenter, randomized, double-blind, parallel-controlled study.

ELIGIBILITY:
Inclusion Criteria:

1. To meet the new diagnosed type 2 diabetes patients, never received oral hypoglycemic drugs or insulin therapy;
2. In accordance with the nonalcoholic fatty liver (NAFLD) criteria for the diagnosis of patients.
3. the level of HbA1c was 7 -10.0%;
4. age 18-70, body mass index 21-35kg/m2;
5. the subjects informed consent and signed the informed consent.

Exclusion Criteria:

1. type 1 diabetes or secondary diabetes;
2. suffering from other liver diseases, such as hepatitis, self - free liver, etc.
3. abnormal thyroid function (in the active period), or the need for long-term oral and intravenous glucocorticoids to treat patients;
4. patients with severe renal dysfunction or renal disease (eGFR<60);
5. in those with abnormal liver function, Alanine transaminase(ALT) or Aspartate transaminase(AST) was more than 3 times the normal upper limit.
6. people with serious gastrointestinal diseases such as peptic ulcers and chronic diarrhea;
7. patients with severe cardiopulmonary disease, cerebrovascular disease or stents;
8. hemopoietic system diseases such as serious primary diseases, hemoglobin < 100g/L or need regular transfusion treatment;
9. pregnant, breast-feeding, women of childbearing age who are unwilling to contraception during the study period;
10. chronic cardiac insufficiency, the classification of heart function III level and above;
11. uncontrolled malignant tumor, and the history of bladder cancer.
12. acute complications of diabetes;
13. the use of other drugs for diabetes and liver disease;
14. patients who had participated in other clinical studies within three months;
15. people who have known allergies to this kind of drugs are known.
16. it is impossible to guarantee the effect or the safety judgment of the drug or the person who is unable to cooperate with the mental illness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-04-28 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Decreased of liver fat content of fatty liver after 24 weeks treatment as assessed by B-ultrasound | up to 24 weeks
  Change from baseline liver fat content to up to 24 weeks after treatment
Change of B-cell function after 24 weeks treatment as assessed by homeostasis model assessment of insulin resistance index | up to 24 weeks
  Change from baseline B-cell function to up to 24 weeks after treatment
Change of liver enzyme after 24 weeks treatment as assessed by blood test | up to 24 weeks
  Change from baseline liver enzyme to up to 24 weeks after treatment

SECONDARY OUTCOMES:
Decreased of HbA1c after 24 weeks treatment as assessed by blood test | up to 24 weeks
  Change from baseline HbA1c to up to 24 weeks after treatment
Decreased of fasting blood glucose after 24 weeks treatment as assessed by blood test | up to 24 weeks
  Change from baseline fasting blood glucose to up to 24 weeks after treatment
Change of weight and waistline after 24 weeks treatment as assessed by standard measurement | up to 24 weeks
  Change from baseline weight and waistline to up to 24 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Qiuhe Ph.D Ji, M.D., Principal Investigator — Department of Endocrinology,Xi jing Hospital,Fourth Military Medical University
Locations (1):
- Xijing Hospital, Fourth Military Medical university, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jianfang F, Wanxia X, Xiling G, Jing X, Wenjuan Y, Jianrong L, Qingzhen H, Kaiyan M, Jingxuan L, Taixiong C, Qian X, Mengying L, Jie M, Qiuhe J. Effect and Safety of Pioglitazone-Metformin Tablets in the Treatment of Newly Diagnosed Type 2 Diabetes Patients with Nonalcoholic Fatty Liver Disease in Shaanxi Province: A Randomized, Double-Blinded, Double-Simulated Multicenter Study. J Diabetes Res. 2023 Jun 1;2023:2044090. doi: 10.1155/2023/2044090. eCollection 2023. PMID 37305429